CLINICAL TRIAL: NCT03787719
Title: Dialysis-Less Frequently In The Elderly (D-LITE) Pilot Study
Brief Title: Dialysis-Less Frequently In The Elderly
Acronym: D-LITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Christine White (Other)
Responsible Party: Sponsor-Investigator, Dr. Christine White, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6021932
Record Dates: First submitted 2018-12-11; First posted 2018-12-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dialysis; End Stage Renal Disease; Hemodialysis
Keywords: Twice weekly dialysis; Thrice weekly dialysis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Single center pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twice per week dialysis (Experimental): Twice-weekly 4 hour dialysis treatment (Monday and Friday or Tuesday and Saturday).
  Interventions: Other: Twice per week dialysis
- Thrice per week dialysis (No Intervention): Standard thrice-weekly 4 hour dialysis treatment (Monday, Wednesday and Friday or Tuesday, Thursday and Staurday)

INTERVENTIONS:
Other: Twice per week dialysis — Twice-weekly 4 hour dialysis treatment
  Arms: Twice per week dialysis

SUMMARY:
Thrice-weekly dialysis is the accepted standard of care for hemodialysis (HD) patients. Observational studies suggest that elderly HD patients do as well and have better quality of life with less dialysis (ie twice-weekly). We propose a single-center pilot study of 40 patients to determine the feasibility of a large randomized controlled trial (RCT) designed to determine the impact of HD frequency on well-being in new HD patients above the age of 70. The primary outcomes will be metrics of feasibility and safety. We hypothesize that an adequately powered RCT that will determine whether elderly patients who dialyze twice weekly have improved well-being compared to thrice-weekly is feasible

DETAILED DESCRIPTION:
This single-center pilot study of 40 patients is designed to determine the feasibility and safety of a large randomized controlled trial examining the impact of hemodialysis frequency on well-being, a patient reported outcome, in incident patients with end stage kidney disease who are above the age of 70. Subjects meeting inclusion criteria will be enrolled into the trial if they are still alive 7 weeks post HD initiation. Once enrolled, subjects will continue thrice weekly HD, have weekly potassium measured, have intra-dialytic weight gain and dry weight assessed weekly and have any extra or missed HD sessions and death recorded. Six weeks post enrollment, subjects meeting inclusion for randomization (potassium within normal range on K2,3 or 4 bath and mean inter-dialytic weight gain of less than 2 L and within 1.0 kg of their prescribed dry weight on weeks 5 and 6) will have residual GFR measured by iohexol clearance and by the average of 48 hour urea and creatinine clearance. Randomization will be 1:1 using permuted blocks of undisclosed varying size and stratified by residual kidney function (RKF) (<5 ml/min, 5-10 ml/min and >10 ml/min) measured by the average of 48 hour urea and creatinine clearance. Throughout the remaining 9 months, potassium will be measured weekly, interdialytic weight gain recorded, and missed or extra HD sessions and death will be recorded. Every 6 weeks, ESAs-r and every 3 months the SF-36 will be completed. The primary outcome for this single-center pilot study will be metrics of feasibility and safety. Feasibility will be assessed by rate of enrollment into the trial and rate of subsequent randomization to a treatment arm, adherence to protocol and loss to trial completion. Safety will be assessed by measures of serum potassium and achievement of target weight. We hypothesize that an adequately powered RCT (The D-LITE Main Trial) that will determine whether elderly patients who dialyze twice weekly have better self-reported well-being compared to thrice weekly will be feasible.

ELIGIBILITY:
Inclusion Criteria:

* Greater than equal 70 years old, planned ongoing in-center HD treatment
* Incident HD patient and still alive 7 weeks post HD initiation
* Patient or substitute decision maker provide informed consent

Exclusion Criteria:

* Significant barriers to ascertainment of the patient-reported experience measures
* Patient currently admitted to hospital without Alternate Level of Care designation
* Patient non-adherent to dialysis prescription

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Recruitment | 1 year
  Successful recruitment will be defined as >3-4 patients/month over 12 months providing informed consent and meeting criteria for randomization.
percent of prescribed treatments completed by patient | 1 year
  Successful adherence will be defined as => 90% of intervention being adhered to.
Loss to trial completion | 1 year
  Successful loss to trial completion will be defined as = >50% of randomized patients completing the 12 month trial. Based on our data, the anticipated reasons for loss to trial completion will be death and moving away from the study center.
Percent of weekly potassium values falling within normal range. | 1 year
  Potassium will be measured every week for the duration of the study.
Percent of weekly post hemodialysis weights that are within 1 kg of prescribed dry weight | 1 year
  Prescribed and acheived post HD weight will be recorded weekly.

SECONDARY OUTCOMES:
Change in Patient's Quality of Life - Using Edmonton Symptom Assessment System (ESAS-R) | 1 year
  The purpose of the ESAS tool is to help with the assessment of 9 symptoms which includes: pain, tiredness, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath and well-being.
  The ESAS-R is a semantic differential scale which asks respondents to answer a questionnaire and choose between two opposite position (e.g., "No Pain" or "Worst Possible Pain", "No Tiredness" or "Worst Possible Tiredness", etc). The patient will rate the severity of each symptom from 0 to 10. The lower the value the better the outcome.
  This study will measure the change in ESAS-r symptoms over time. The ESAS-r is always done on the ESAS-r numerical scale and the results later transferred to the ESAS-r Graph.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre (KHSC), Kingston, Ontario, Canada